CLINICAL TRIAL: NCT01398800
Title: Early Clinical Results of Mobile-Bearing Revision Total Knee Arthroplasty
Acronym: MBT
Status: Completed | Type: Observational
Sponsor: Colorado Joint Replacement (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Donnis Rafferty, Dr. Raymond Kim, Colorado Joint Replacement
Other Study IDs: IIS-000113
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Long term follow-up is needed to determine whether current Mobile Bearing revision Total Knee Arthroplasty (TKA) designs will improve implant longevity. The potential advantages of mobile bearings in the revision TKA setting include reduction in polyethylene wear, decreasing fixation stresses, and protection of the constraining mechanisms. Several studies have reported satisfactory clinical results after revision total knee arthroplasty but no study with a large number has specifically addressed the clinical outcomes after revision total knee arthroplasty using the mobile bearing design

DETAILED DESCRIPTION:
Failure modes of revision total knee arthroplasty (TKA) that include prosthetic loosening and damage to constraining mechanisms often require revision TKA. Mobile bearing revision TKA components have been developed in hopes of lessening these failure mechanisms. Our purpose is to evaluate the use of mobile bearings in revision TKA.

Retrospective clinical and radiographic evaluation of 340 revision mobile bearing TKAs using the PFC Sigma and LCS posterior stabilized rotating platform implants (Depuy, Warsaw, IN) will be performed. Indications for revision include instability, loosening, arthrofibrosis, chronic hemarthrosis, failed patellofemoral replacement, failed unicompartmental knee replacement, infection reimplantation, and supracondylar fracture nonunion.

ELIGIBILITY:
Inclusion Criteria:

Requiring a revision of a primary knee replacement. Indications for revision include instability, aseptic loosening, failed unicompartmental knee replacement, infection reimplantation, arthrofibroisis, chronic hemarthrosis, failed patellofemoral replacments, and non union of a supracondylar femur fracture.

Exclusion Criteria: None since they have all required a revision.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients of Colorado Joint Replacement
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2011-07; Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Function and knee score of the knee society scoring at every 2 years until 10 years. | 1-10 years post operative of revision
  Follow up data of 1,2,4,6,8,and 10 years to evaluate bearing complications and clinical results for the use of MB in revision TKA. Retrospective clinical and radiographic evaluation of 197 mobile bearing revision TKA's will be collected. We will also analyze patient demographics and reason for revisions as well as implants used in revision.

SECONDARY OUTCOMES:
Radiographic analysis by our orthopedic clinician to determine component failure or loosening. | Post op - 1-10 years or revision surgery

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kim, MD, Principal Investigator — Colorado Joint Replacement
Locations (1):
- Colorado Joint Replacement, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided